CLINICAL TRIAL: NCT07401628
Title: Randomised, Controlled, Interventional Single-center Study for the Design and Evaluation of an In-vehicle Real-time System for Detecting Cannabis-impaired Driving (CID)
Brief Title: In-Vehicle Real-Time Cannabis Influenced Driving Detection
Acronym: REVELIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: ETH Zurich (Other); University of St.Gallen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-01590
Record Dates: First submitted 2026-01-22; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Driving Under the Influence; Cannabis-impaired Driving
MeSH Terms: conditions — Driving Under the Influence | interventions — nabiximols; Dronabinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controlled Cannabis Administration (Experimental): Participants assigned to this arm receive a single, controlled inhalative administration of cannabis by smoking a THC-containing joint with a target dose of approximately 0.67 mg THC per kg body weight. Participants complete standardized driving sessions in an instrumented vehicle on a closed test track under sober baseline conditions and repeatedly after cannabis administration (approximately 1-6 hours post-dose). All driving sessions are conducted with a certified driving instructor seated in the front passenger seat with access to dual pedals, allowing immediate intervention if required. Multimodal in-vehicle sensor data, physiological signals, driving performance measures, and biological samples are collected throughout the study.
  Interventions: Drug: Cannabis (THC)
- Reference (No Cannabis) (No Intervention): Participants assigned to this reference arm receive no cannabis administration. They complete the same screening procedures, standardized driving sessions, assessments, and data collection as the experimental group under sober conditions, following the same schedule and time points. All driving sessions are conducted with a certified driving instructor seated in the front passenger seat with access to dual pedals, ensuring identical safety conditions. This arm serves as a non-impaired reference for comparison of driving behavior and in-vehicle sensor data.

INTERVENTIONS:
Drug: Cannabis (THC) — Participants assigned to the experimental arm receive a single, controlled inhalative administration of cannabis by smoking a THC-containing joint (target dose 0.67 mg THC per kg body weight; cannabis flowers with 15-18% THC).
  Arms: Controlled Cannabis Administration

SUMMARY:
The goal of this clinical trial is to evaluate whether in-vehicle sensor data can be used to detect cannabis-impaired driving in healthy adult recreational cannabis users.

The study aims to assess whether changes in vehicle, driver, and physiological sensor data can distinguish sober driving from cannabis-impaired driving, and how driving performance changes from baseline to approximately 1 to 6 hours after controlled cannabis consumption.

Researchers will compare driving behavior and in-vehicle sensor data from participants who receive controlled cannabis administration with data from a randomized reference group without cannabis exposure, to determine whether cannabis-related impairment driving can be identified on the basis of machine learning.

Participants will complete screening and baseline assessments and drive an instrumented vehicle on a closed test track under sober conditions. Participants assigned to the experimental arm will receive controlled cannabis administration, while participants in the reference arm will receive no intervention. All participants will perform repeated standardized driving sessions over several hours and complete traffic-medical, traffic-psychological, and in-vehicle pre-driving tests. Biological samples and in-vehicle sensor data will be collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Recreational cannabis-consumption (more than once per month)
* In possession of a definite Swiss or European Union (EU) driving license
* At least 21 years old
* Active, regular driving a car in the last 6 months
* Must be in good health condition
* No special equipment needed when driving (special seats, levers, etc.)
* Fluent in (Swiss) German and no speech impairment

Exclusion Criteria:

* Health concerns where cannabis consumption is contra-indicated (such as: high blood pressure, psychiatric problems (e.g. psychosis, depression, attention-deficit conditions, etc.)
* Cannabis-abstinence or excessive consumption, , assessed using the Cannabis Use Disorders Identification Test-Revised (CUDIT-R)
* For women: pregnancy or breastfeeding or if intention to become pregnant during study period (time between telephone screening and study day (visit 2)
* Alcohol misuse or excessive alcohol consumption habits/risky drinking behaviour, assessed using the Alcohol Use Disorders Identification Test (AUDIT) and/or phosphatidylethanol (PEth) in capillary blood > 200 ng/mL at first visit
* If breath alcohol test is positive at Visit 1 or Visit 2 (study day)
* Consumption of drugs of abuse (others than cannabis) within 4 weeks before the study
* Consumption of medications / pharmaceutical drugs which interfere with driving ability
* Inability to follow the procedures of the study, e.g., due to language

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnancy test is required for females
Enrollment: 45 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-06-19 (Estimated); Study Completion 2026-06-19 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy (AUROC) of a multimodal machine-learning model for detection of cannabis-impaired driving | Baseline (sober driving) and up to 6 hours after cannabis administration in the experimental arm, with matched time points in the reference arm.
  Area under the receiver operating characteristic curve (AUROC) of a single machine-learning classifier that integrates multimodal in-vehicle data (including vehicle controller area network [CAN] data, driver monitoring camera [DMC] features, and physiological signals). All modalities are combined into one predictive model, and performance is reported as one aggregated AUROC value distinguishing non-impaired (sober) driving from cannabis-impaired driving.

SECONDARY OUTCOMES:
Diagnostic accuracy (AUROC) using CAN data | Baseline (sober driving) and approximately 1-2, 3-4, and 5-6 hours after cannabis administration in the experimental arm, with matched time points in the reference arm.
  AUROC for detecting cannabis-impaired driving using vehicle controller area network (CAN) data only.
Diagnostic accuracy (AUROC) using DMC data | Baseline (sober driving) and approximately 1-2, 3-4, and 5-6 hours after cannabis administration in the experimental arm, with matched time points in the reference arm.
  AUROC for detecting cannabis-impaired driving using driver monitoring camera (DMC) data only.
Diagnostic accuracy (AUROC) of a physiology-based machine-learning model for detection of cannabis-impaired driving | Baseline (sober driving) and approximately 1-2, 3-4, and 5-6 hours after cannabis administration in the experimental arm, with matched time points in the reference arm.
  AUROC of a single machine-learning classifier trained and evaluated using aggregated physiological features only, derived from signals including heart rate, heart-rate variability, oxygen saturation, electrodermal activity, skin temperature, and respiration-related measures. All physiological signals are combined into one predictive model, and performance is reported as a single AUROC value distinguishing non-impaired (sober) driving from cannabis-impaired driving.
Change in driving behavior derived from vehicle CAN data | Baseline (sober driving) and approximately 1-2, 3-4, and 5-6 hours after cannabis administration in the experimental arm, with matched time points in the reference arm.
  Change in driving behavior between sober driving and post-cannabis driving, derived from vehicle controller area network (CAN) signals, including steering, braking, acceleration, and velocity-related measures.
Change in driver gaze behavior derived from DMC data | Baseline (sober driving) and approximately 1-2, 3-4, and 5-6 hours after cannabis administration in the experimental arm, with matched time points in the reference arm.
  Change in gaze behavior between sober and post-cannabis driving, derived from driver monitoring camera (DMC) data, including gaze direction and gaze dynamics during driving.
Change in head movement behavior derived from DMC data | Baseline (sober driving) and approximately 1-2, 3-4, and 5-6 hours after cannabis administration in the experimental arm, with matched time points in the reference arm.
  Change in head movement behavior between sober and post-cannabis driving, derived from driver monitoring camera (DMC) data.
Driving instructor assessment of driving performance | Baseline (sober driving) and approximately 1-2, 3-4, and 5-6 hours after cannabis administration in the experimental arm, with matched time points in the reference arm.
  Assessment of driving performance conducted by a certified driving instructor, quantified as the number of safety interventions required during each standardized driving session.
Diagnostic accuracy (AUROC) of an in-vehicle pre-driving readiness test for detection of cannabis-impaired driving | Baseline (sober driving) and approximately 1-2, 3-4, and 5-6 hours after cannabis administration in the experimental arm, with matched time points in the reference arm.
  AUROC of a machine-learning (ML) classification model implementing a study-specific in-vehicle pre-driving readiness test. The test produces an ML-derived readiness score, computed from features derived from the pre-driving test (e.g., attention-related, reaction-time-related, and psychomotor-related features), and is used to classify driving sessions as sober versus post-cannabis.
Performance in the standardized Psytest assessment | Baseline (sober driving) and approximately 1-2, 3-4, and 5-6 hours after cannabis administration in the experimental arm, with matched time points in the reference arm.
  Performance in the standardized Psytest assessment (mobility version of the Test of Attentional Performance), administered under sober conditions and after cannabis consumption. Test performance is summarized using a standardized test score reflecting overall attentional and psychomotor performance relevant for driving.
Self-reported subjective effects | Baseline (sober driving) and approximately 1-2, 3-4, and 5-6 hours after cannabis administration in the experimental arm, with matched time points in the reference arm.
  Self-reported subjective effects assessed using study questionnaires, including subjective feeling of "high" and degree of sleepiness. Responses are recorded using a Likert scale ranging from 0 to 10, where 0 indicates "not at all" and 10 indicates "extremely." Higher scores indicate a worse outcome, reflecting stronger subjective drug effects and greater sleepiness.
Cannabinoid biomarker concentrations in biological samples | Baseline in all participants, and approximately 1-2, 3-4, and 5-6 hours after cannabis administration in the experimental arm.
  Concentrations of Δ9-tetrahydrocannabinol (THC) measured in capillary blood, oral fluid, and breath samples.
Incidence of adverse events | From the first study procedure (i.e. baseline assessment) to the end of the main study day (i.e. driving assessment) expected to be on average up to 6 hours.
  Incidence of adverse events and serious adverse events recorded during all study visits.
Change in heart rate during driving | Baseline (sober driving) and approximately 1-2, 3-4, and 5-6 hours after cannabis administration in the experimental arm, with matched time points in the reference arm.
  Change in heart rate measured during driving between sober conditions and post-cannabis conditions.
Change in oxygen saturation during driving | Baseline (sober driving) and approximately 1-2, 3-4, and 5-6 hours after cannabis administration in the experimental arm, with matched time points in the reference arm.
  Change in oxygen saturation measured during driving between sober conditions and post-cannabis conditions.
Change in electrodermal activity during driving | Baseline (sober driving) and approximately 1-2, 3-4, and 5-6 hours after cannabis administration in the experimental arm, with matched time points in the reference arm.
  Change in electrodermal activity measured during driving between sober conditions and post-cannabis conditions.
Change in skin temperature during driving | Baseline (sober driving) and approximately 1-2, 3-4, and 5-6 hours after cannabis administration in the experimental arm, with matched time points in the reference arm.
  Change in skin temperature measured during driving between sober conditions and post-cannabis conditions.
Change in respiration during driving | Baseline (sober driving) and approximately 1-2, 3-4, and 5-6 hours after cannabis administration in the experimental arm, with matched time points in the reference arm.
  Change in respiration measured during driving between sober conditions and post-cannabis conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Weinmann, Prof. Dr., Principal Investigator — Institute for Forensic Medicine, Forensic Chemistry and Toxicology University of Bern
Locations (1):
- Institute for Forensic Medicine, Forensic Chemistry and Toxicology University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No